CLINICAL TRIAL: NCT06781801
Title: Longitudinal Approach to Generate Positive Cardiometabolic Health Outcomes in Severe Mental Illness
Brief Title: Improving Heart and Metabolic Health in People With Severe Mental Illness Through a Long-term Clinical Trial
Acronym: LAGOM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: The Swedish Society of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CIV-24-09-049056
Record Dates: First submitted 2025-01-02; First posted 2025-01-17 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-10

CONDITIONS: Psychotic Disorders
Keywords: Psychotic disorders; Quality of life; Cost-effectiveness; Cardiometabolic risk factors; Cardiovascular disease prevention; Metabolic syndrome; Pragmatic clinical trial; Integrated health care; Multicomponent intervention; Behavior change intervention
MeSH Terms: conditions — Psychotic Disorders; Metabolic Syndrome | interventions — Methods

STUDY DESIGN:
Intervention Model Description: This is a longitudinal, multicenter, naturalistic, multicomponent, parallel-group, quasi-experimental cluster-based trial with a superiority framework. The trial uses a case-control clinical design with a 1:3 allocation ratio, assigning one participant at the intervention clinics for every three at the control clinics. Clusters are defined at the level of outpatient clinics, with two intervention clinics and four control clinics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control clinics (usual care) (No Intervention): The "usual care" model in Gothenburg includes annual health checks for individuals with psychotic disorders. Patients attend two 60-minute visits for assessments such as blood tests, blood pressure, and weight checks, with results evaluated using standard benchmarks or risk algorithms like SCORE2. Physicians may suggest referrals to primary care or recommend lifestyle changes, including diet, exercise, or substance use adjustments. Identified issues may prompt simple advice or referrals to health promoters for support with smoking cessation, dietary guidance, or group activities.
  The 36 ± 6-month clinical trial standardizes data collection at four outpatient clinics without altering care. Eligible patients sign consent, with rescreening allowed if a patient meets the exclusion criteria at one annual check but not at the next. Non-participants continue with regular care.
- Intervention Clinics (Experimental): The annual health checks for the intervention group follow the same structure of two visits as in routine care as usual, with the primary difference being the content of the visits.
  Interventions: Other: Intervention

INTERVENTIONS:
Other: Intervention — The intervention group follows a structured flowchart for annual health check-ups, focusing on assessing the cardiometabolic profile, considering sex and ethnicity. This assessment includes tracking changes in cardiometabolic parameters, alongside overall cardiometabolic risk using SCORE2 and if the criteria for metabolic syndrome are met.
  Lifestyle habits are evaluated based on health status, illness, and benefits of quitting unhealthy behaviors. Education sessions educate participants and families on the link between psychotic disorders, lifestyle choices, and cardiometabolic health.
  Gradual lifestyle changes are tailored to individual needs, addressing stress and cognitive challenges, and follow national health guidelines with personalized advice and motivational tools. Regular follow-ups assess progress, while motivational tools "body composition analyzer and QRISK3" enhance engagement. Contact with internal and external resources is based on the assessment and motivational work.
  Arms: Intervention Clinics

SUMMARY:
Cardiometabolic diseases are prevalent among individuals with psychotic disorders, significantly contributing to their shorter lifespan, reduced quality of life, and economic impact on individuals and society. To improve cardiometabolic health, effective and individualized interventions are crucial. Psychosis outpatient clinics are ideal for these interventions due to regular patient visits and the availability of diverse health professionals. The investigators have developed and want to test a comprehensive intervention program to improve cardiometabolic health, enhance quality of life, and promote healthy lifestyles specifically for people with psychotic disorders at psychiatric outpatient clinics in Gothenburg.

This clinical trial aims to include 644 individuals with psychotic disorders from six outpatient clinics in the Department of Psychotic Disorders at Sahlgrenska University Hospital in Gothenburg. Two outpatient clinics will provide the LAGOM-intervention, while the other clinics will serve as controls, offering "care as usual". The intervention group will receive multidisciplinary support integrated into the routine clinical procedures. The intervention includes regular follow-ups and use of motivational tools, including body composition analyzer and cardiovascular risk prediction algorithm (QRISK3).

If the intervention effectively improves cardiometabolic health, enhances quality of life for this vulnerable group, and proves cost-effective, it can serve as a model program for implementation in Region Västra Götaland.

ELIGIBILITY:
Inclusion criteria

1. Adults ≥18 years of age meeting the International Classification of Diseases, Tenth Revision (ICD-10) diagnostic criteria for any one of the schizophrenia spectrum disorders (F20-F25 or F28-F29)
2. Ability to provide informed consent

Exclusion criteria

1. Having an electrical medical implant such as a pacemaker or other mechanical implants
2. Pregnancy
3. Deemed unsuitable by the investigator (a person may be deemed unsuitable for participation in the trial by the clinical investigation team member based on factors that may affect the ability to participate safely and reliably. These factors may include, but are not limited to, physical disabilities that hinder participation or practical challenges such as long travel distances to the trial site. The assessment is made on an individual basis and aims to ensure both patient safety and trial integrity).
4. Prior participation in the LAGOM trial during a previous inclusion cycle (i.e., participants can only be included once during the trial period).
5. Currently under compulsory care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 644 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in body mass index | At 12 months from baseline.
  To evaluate whether the intervention is superior to usual care in reducing cardiometabolic risk indicators over the 36-month period.
  Primary endpoint:
  Differences in the mean changes in body mass index (BMI) (kg/m2).
Change in body mass index | At 24 months from baseline.
  To evaluate whether the intervention is superior to usual care in reducing cardiometabolic risk indicators over the 36-month period.
  Primary endpoint:
  Differences in the mean changes in body mass index (BMI) (kg/m2).
Change in body mass index | At 36 months from baseline.
  To evaluate whether the intervention is superior to usual care in reducing cardiometabolic risk indicators over the 36-month period.
  Primary endpoint:
  Differences in the mean changes in body mass index (BMI) (kg/m2).
Change in waist-hip ratio | At 12 months from baseline.
  To evaluate whether the intervention is superior to usual care in reducing cardiometabolic risk indicators over the 36-month period.
  Primary endpoint:
  Differences in the mean changes in waist-hip ratio (WHR).
Change in waist-hip ratio | At 24 months from baseline.
  To evaluate whether the intervention is superior to usual care in reducing cardiometabolic risk indicators over the 36-month period.
  Primary endpoint:
  Differences in the mean changes in waist-hip ratio (WHR).
Change in waist-hip ratio | At 36 months from baseline.
  To evaluate whether the intervention is superior to usual care in reducing cardiometabolic risk indicators over the 36-month period.
  Primary endpoint:
  Differences in the mean changes in waist-hip ratio (WHR).
Change in systolic blood pressure | At 12 months from baseline.
  To evaluate whether the intervention is superior to usual care in reducing cardiometabolic risk indicators over the 36-month period.
  Primary endpoint:
  Differences in the mean changes in systolic blood pressure (SBP) (mm Hg).
Change in systolic blood pressure | At 24 months from baseline.
  To evaluate whether the intervention is superior to usual care in reducing cardiometabolic risk indicators over the 36-month period.
  Primary endpoint:
  Differences in the mean changes in systolic blood pressure (SBP) (mm Hg).
Change in systolic blood pressure | At 36 months from baseline.
  To evaluate whether the intervention is superior to usual care in reducing cardiometabolic risk indicators over the 36-month period.
  Primary endpoint:
  Differences in the mean changes in systolic blood pressure (SBP) (mm Hg).
Change in diastolic blood pressure | At 12 months from baseline.
  To evaluate whether the intervention is superior to usual care in reducing cardiometabolic risk indicators over the 36-month period.
  Primary endpoint:
  Differences in the mean changes in diastolic blood pressure (DBP) mm Hg.
Change in diastolic blood pressure | At 24 months from baseline.
  To evaluate whether the intervention is superior to usual care in reducing cardiometabolic risk indicators over the 36-month period.
  Primary endpoint:
  Differences in the mean changes in diastolic blood pressure (DBP) mm Hg.
Change in diastolic blood pressure | At 36 months from baseline.
  To evaluate whether the intervention is superior to usual care in reducing cardiometabolic risk indicators over the 36-month period.
  Primary endpoint:
  Differences in the mean changes in diastolic blood pressure (DBP) mm Hg.
Change in triacylglycerol/high density lipoprotein-cholesterol ratio | At 12 months from baseline.
  To evaluate whether the intervention is superior to usual care in reducing cardiometabolic risk indicators over the 36-month period.
  Primary endpoint:
  Differences in the mean changes in triacylglycerol/high density lipoprotein-cholesterol ratio (TAG/HDL-C ratio).
Change in triacylglycerol/high density lipoprotein-cholesterol ratio | At 24 months from baseline.
  To evaluate whether the intervention is superior to usual care in reducing cardiometabolic risk indicators over the 36-month period.
  Primary endpoint:
  Differences in the mean changes in triacylglycerol/high density lipoprotein-cholesterol ratio (TAG/HDL-C ratio).
Change in triacylglycerol/high density lipoprotein-cholesterol ratio | At 36 months from baseline.
  To evaluate whether the intervention is superior to usual care in reducing cardiometabolic risk indicators over the 36-month period.
  Primary endpoint:
  Differences in the mean changes in triacylglycerol/high density lipoprotein-cholesterol ratio (TAG/HDL-C ratio).
Change in total cholesterol/HDL-C ratio | At 12 months from baseline.
  To evaluate whether the intervention is superior to usual care in reducing cardiometabolic risk indicators over the 36-month period.
  Primary endpoint:
  Differences in the mean changes in total cholesterol/HDL-C ratio (TChol/HDL-C ratio).
Change in total cholesterol/HDL-C ratio | At 24 months from baseline.
  To evaluate whether the intervention is superior to usual care in reducing cardiometabolic risk indicators over the 36-month period.
  Primary endpoint:
  Differences in the mean changes in total cholesterol/HDL-C ratio (TChol/HDL-C ratio).
Change in total cholesterol/HDL-C ratio | At 36 months from baseline.
  To evaluate whether the intervention is superior to usual care in reducing cardiometabolic risk indicators over the 36-month period.
  Primary endpoint:
  Differences in the mean changes in total cholesterol/HDL-C ratio (TChol/HDL-C ratio).
Change in plasma glucose | At 12 months from baseline.
  To evaluate whether the intervention is superior to usual care in reducing cardiometabolic risk indicators over the 36-month period.
  Primary endpoint:
  Differences in the mean changes in plasma glucose (mmol/L).
Change in plasma glucose | At 24 months from baseline.
  To evaluate whether the intervention is superior to usual care in reducing cardiometabolic risk indicators over the 36-month period.
  Primary endpoint:
  Differences in the mean changes in plasma glucose (mmol/L).
Change in plasma glucose | At 36 months from baseline.
  To evaluate whether the intervention is superior to usual care in reducing cardiometabolic risk indicators over the 36-month period.
  Primary endpoint:
  Differences in the mean changes in plasma glucose (mmol/L).

SECONDARY OUTCOMES:
Change in cardiovascular disease (CVD) events or risk scores based on the SCORE2 algorithm | At 36 months from baseline.
  To assess whether the intervention is superior to usual care in reducing the risk of cardiovascular disease (CVD) at 36 months.
  Secondary endpoint:
  CVD outcomes: Hazard ratio of incident CVD events and/or differences in the mean change in the CVD risk score will be assessed using the Systematic COronary Risk Evaluation 2 (SCORE2), a tool designed to estimate the 10-year risk of cardiovascular events in individuals aged 40-89 years. SCORE2 ranges from a minimum value of 0% (indicating no risk) to a maximum value of 100% (indicating certainty of an event). Higher scores represent a worse outcome, as they reflect an increased likelihood of experiencing a cardiovascular event within the specified timeframe.
Change in incident rate of type 2 diabetes mellitus events | At 36 months from baseline.
  To assess whether the intervention is superior to usual care in reducing type 2 diabetes mellitus at 36 months.
  Secondary endpoints:
  Diabetes mellitus outcomes: Hazard ratio of incident type 2 diabetes mellitus events.

OTHER OUTCOMES:
Change in quality of life | At 12 months from baseline.
  To evaluate whether the intervention is superior to usual care in improving health-related quality of life over the 36-month period.
  Other endpoint:
  Difference in the mean change in the quality of life questionnaire (EQ-5D-5L)*.
  *Quality of life according to the EuroQol 5-Dimension 5-Level (EQ-5D-5L) Questionnaire, which measures five dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Respondents indicate problems on each dimension at one of five levels: no problems, slight problems, moderate problems, severe problems, or extreme problems/unable to perform. The EQ-5D-5L classification system can describe 3,125 possible health states. Additionally, the EQ-5D-5L includes a visual analogue scale (EQ VAS), where respondents rate their current health on a scale from 0 (the worst health they can imagine) to 100 (the best health they can imagine).
Change in quality of life | At 24 months from baseline.
  To evaluate whether the intervention is superior to usual care in improving health-related quality of life over the 36-month period.
  Other endpoint:
  Difference in the mean change in the quality of life questionnaire (EQ-5D-5L)*.
  *Quality of life according to the EuroQol 5-Dimension 5-Level (EQ-5D-5L) Questionnaire, which measures five dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Respondents indicate problems on each dimension at one of five levels: no problems, slight problems, moderate problems, severe problems, or extreme problems/unable to perform. The EQ-5D-5L classification system can describe 3,125 possible health states. Additionally, the EQ-5D-5L includes a visual analogue scale (EQ VAS), where respondents rate their current health on a scale from 0 (the worst health they can imagine) to 100 (the best health they can imagine).
Change in quality of life | At 36 months from baseline.
  To evaluate whether the intervention is superior to usual care in improving health-related quality of life over the 36-month period.
  Other endpoint:
  Difference in the mean change in the quality of life questionnaire (EQ-5D-5L)*.
  *Quality of life according to the EuroQol 5-Dimension 5-Level (EQ-5D-5L) Questionnaire, which measures five dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Respondents indicate problems on each dimension at one of five levels: no problems, slight problems, moderate problems, severe problems, or extreme problems/unable to perform. The EQ-5D-5L classification system can describe 3,125 possible health states. Additionally, the EQ-5D-5L includes a visual analogue scale (EQ VAS), where respondents rate their current health on a scale from 0 (the worst health they can imagine) to 100 (the best health they can imagine).
Change in high-sensitivity C-reactive protein | At 12 months from baseline.
  To assess whether the intervention reduces the levels of high-sensitivity C-reactive protein (hs-CRP) over the 36-month period.
  Other endpoints:
  Differences in the mean changes in hs-CRP (mg/L).
Change in high-sensitivity C-reactive protein | At 24 months from baseline.
  To assess whether the intervention reduces the levels of high-sensitivity C-reactive protein (hs-CRP) over the 36-month period.
  Other endpoints:
  Differences in the mean changes in hs-CRP (mg/L).
Change in high-sensitivity C-reactive protein | At 36 months from baseline.
  To assess whether the intervention reduces the levels of high-sensitivity C-reactive protein (hs-CRP) over the 36-month period.
  Other endpoints:
  Differences in the mean changes in hs-CRP (mg/L).
Change in HbA1c | At 12 months from baseline.
  To assess whether the intervention reduces the levels of HbA1c over the 36-month period.
  Other endpoints:
  Differences in the mean changes in HbA1c (mmol/mol).
Change in HbA1c | At 24 months from baseline.
  To assess whether the intervention reduces the levels of HbA1c over the 36-month period.
  Other endpoints:
  Differences in the mean changes in HbA1c (mmol/mol).
Change in HbA1c | At 36 months from baseline.
  To assess whether the intervention reduces the levels of HbA1c over the 36-month period.
  Other endpoints:
  Differences in the mean changes in HbA1c (mmol/mol).
Descriptive cost analysis | At 12 months from baseline.
  To conduct a cost analysis per participant and assess cost-effectiveness over the 36-month period, where cost neutrality is considered a positive outcome.
  Other endpoint:
  Descriptive cost analysis (average cost per participant) in SEK and EUR.
Descriptive cost analysis | At 24 months from baseline.
  To conduct a cost analysis per participant and assess cost-effectiveness over the 36-month period, where cost neutrality is considered a positive outcome.
  Other endpoint:
  Descriptive cost analysis (average cost per participant) in SEK and EUR.
Descriptive cost analysis | At 36 months from baseline.
  To conduct a cost analysis per participant and assess cost-effectiveness over the 36-month period, where cost neutrality is considered a positive outcome.
  Other endpoint:
  Descriptive cost analysis (average cost per participant) in SEK and EUR.
Change in quality-Adjusted Life Years | At 12 months from baseline.
  To conduct a cost analysis per participant and assess cost-effectiveness over the 36-month period, where cost neutrality is considered a positive outcome.
  Other endpoints:
  Difference in the mean change in quality-adjusted life years (QALYs) between the intervention and control groups.
Change in quality-Adjusted Life Years | At 24 months from baseline.
  To conduct a cost analysis per participant and assess cost-effectiveness over the 36-month period, where cost neutrality is considered a positive outcome.
  Other endpoints:
  Difference in the mean change in quality-adjusted life years (QALYs) between the intervention and control groups.
Change in quality-Adjusted Life Years | At 36 months from baseline.
  To conduct a cost analysis per participant and assess cost-effectiveness over the 36-month period, where cost neutrality is considered a positive outcome.
  Other endpoints:
  Difference in the mean change in quality-adjusted life years (QALYs) between the intervention and control groups
Incremental cost-effectiveness ratio based on CVD | At 12 months from baseline.
  To conduct a cost analysis per participant and assess cost-effectiveness over the 36-month period, where cost neutrality is considered a positive outcome
  Other endpoints:
  Incremental cost-effectiveness ratio (ICER) based on the number of CVD cases averted.
Incremental cost-effectiveness ratio based on CVD | At 24 months from baseline.
  To conduct a cost analysis per participant and assess cost-effectiveness over the 36-month period, where cost neutrality is considered a positive outcome
  Other endpoints:
  Incremental cost-effectiveness ratio (ICER) based on the number of CVD cases averted.
Incremental cost-effectiveness ratio based on CVD | At 36 months from baseline.
  To conduct a cost analysis per participant and assess cost-effectiveness over the 36-month period, where cost neutrality is considered a positive outcome
  Other endpoints:
  Incremental cost-effectiveness ratio (ICER) based on the number of CVD cases averted.
Incremental cost-effectiveness ratio based on type 2 diabetes mellitus | At 12 months from baseline.
  To conduct a cost analysis per participant and assess cost-effectiveness over the 36-month period, where cost neutrality is considered a positive outcome
  Other endpoints:
  Incremental cost-effectiveness ratio (ICER) based on the number of type 2 diabetes mellitus cases averted.
Incremental cost-effectiveness ratio based on type 2 diabetes mellitus | At 24 months from baseline.
  To conduct a cost analysis per participant and assess cost-effectiveness over the 36-month period, where cost neutrality is considered a positive outcome
  Other endpoints:
  Incremental cost-effectiveness ratio (ICER) based on the number of type 2 diabetes mellitus cases averted.
Incremental cost-effectiveness ratio based on type 2 diabetes mellitus | At 36 months from baseline.
  To conduct a cost analysis per participant and assess cost-effectiveness over the 36-month period, where cost neutrality is considered a positive outcome
  Other endpoints:
  Incremental cost-effectiveness ratio (ICER) based on the number of type 2 diabetes mellitus cases averted.
Incremental cost-effectiveness ratio based on QALYs | At 12 months from baseline.
  To conduct a cost analysis per participant and assess cost-effectiveness over the 36-month period, where cost neutrality is considered a positive outcome
  Other endpoints:
  Incremental cost-effectiveness ratio (ICER) based on the number of QALYs gained.
Incremental cost-effectiveness ratio based on QALYs | At 24 months from baseline.
  To conduct a cost analysis per participant and assess cost-effectiveness over the 36-month period, where cost neutrality is considered a positive outcome
  Other endpoints:
  Incremental cost-effectiveness ratio (ICER) based on the number of QALYs gained.
Incremental cost-effectiveness ratio based on QALYs | At 36 months from baseline.
  To conduct a cost analysis per participant and assess cost-effectiveness over the 36-month period, where cost neutrality is considered a positive outcome
  Other endpoints:
  Incremental cost-effectiveness ratio (ICER) based on the number of QALYs gained.
Change in alcohol consumption | At 12 months from baseline.
  To evaluate whether the intervention improves targeted lifestyle behaviors (tobacco smoking, alcohol consumption, physical activity, and dietary habits) over the 36-month period.
  Other endpoints:
  Difference in the mean change in alcohol consumption (Alcohol Use Disorders Identification Test - Consumption (AUDIT-C)*, scale 0-12).
  *The AUDIT-C (Alcohol Use Disorders Identification Test-Consumption) is a brief screening tool consisting of three questions, with scores ranging from 0 to 12 points, used to identify risky alcohol use and potential alcohol use disorders.
Change in alcohol consumption | At 24 months from baseline.
  To evaluate whether the intervention improves targeted lifestyle behaviors (tobacco smoking, alcohol consumption, physical activity, and dietary habits) over the 36-month period.
  Other endpoints:
  Difference in the mean change in alcohol consumption (Alcohol Use Disorders Identification Test - Consumption (AUDIT-C)*, scale 0-12).
  *The AUDIT-C (Alcohol Use Disorders Identification Test-Consumption) is a brief screening tool consisting of three questions, with scores ranging from 0 to 12 points, used to identify risky alcohol use and potential alcohol use disorders.
Change in alcohol consumption | At 36 months from baseline.
  To evaluate whether the intervention improves targeted lifestyle behaviors (tobacco smoking, alcohol consumption, physical activity, and dietary habits) over the 36-month period.
  Other endpoints:
  Difference in the mean change in alcohol consumption (Alcohol Use Disorders Identification Test - Consumption (AUDIT-C)*, scale 0-12).
  *The AUDIT-C (Alcohol Use Disorders Identification Test-Consumption) is a brief screening tool consisting of three questions, with scores ranging from 0 to 12 points, used to identify risky alcohol use and potential alcohol use disorders.
Change in tobacco smoking | At 12 months from baseline.
  To evaluate whether the intervention improves targeted lifestyle behaviors (tobacco smoking, alcohol consumption, physical activity, and dietary habits) over the 36-month period.
  Other endpoints:
  • Questionnaires Difference in the mean change in tobacco smoking* per week.
  *The tobacco smoking questionnaire assesses smoking behavior with targeted questions addressing current smoking status, past smoking history, age at smoking initiation or cessation, and smoking frequency (daily or weekly cigarette consumption).
  For smoking frequency:
  Daily smoking frequency: Minimum = 0 cigarettes/day; Maximum = unlimited (as self-reported by participants).
  Weekly smoking frequency: Minimum = 0 cigarettes/week; Maximum = unlimited (as self-reported by participants).
  Higher values for daily or weekly smoking frequency indicate worse outcomes (greater tobacco use).
Change in tobacco smoking | At 24 months from baseline.
  To evaluate whether the intervention improves targeted lifestyle behaviors (tobacco smoking, alcohol consumption, physical activity, and dietary habits) over the 36-month period.
  Other endpoints:
  • Questionnaires Difference in the mean change in tobacco smoking* per week.
  *The tobacco smoking questionnaire assesses smoking behavior with targeted questions addressing current smoking status, past smoking history, age at smoking initiation or cessation, and smoking frequency (daily or weekly cigarette consumption).
  For smoking frequency:
  Daily smoking frequency: Minimum = 0 cigarettes/day; Maximum = unlimited (as self-reported by participants).
  Weekly smoking frequency: Minimum = 0 cigarettes/week; Maximum = unlimited (as self-reported by participants).
  Higher values for daily or weekly smoking frequency indicate worse outcomes (greater tobacco use).
Change in tobacco smoking | At 36 months from baseline.
  To evaluate whether the intervention improves targeted lifestyle behaviors (tobacco smoking, alcohol consumption, physical activity, and dietary habits) over the 36-month period.
  Other endpoints:
  • Questionnaires Difference in the mean change in tobacco smoking* per week.
  *The tobacco smoking questionnaire assesses smoking behavior with targeted questions addressing current smoking status, past smoking history, age at smoking initiation or cessation, and smoking frequency (daily or weekly cigarette consumption).
  For smoking frequency:
  Daily smoking frequency: Minimum = 0 cigarettes/day; Maximum = unlimited (as self-reported by participants).
  Weekly smoking frequency: Minimum = 0 cigarettes/week; Maximum = unlimited (as self-reported by participants).
  Higher values for daily or weekly smoking frequency indicate worse outcomes (greater tobacco use).
Change in dietary habits | At 12 months from baseline.
  To evaluate whether the intervention improves targeted lifestyle behaviors (tobacco smoking, alcohol consumption, physical activity, and dietary habits) over the 36-month period.
  Other endpoints:
  • Questionnaires Difference in the mean change in dietary habits (dietary index)* (scale 0-12).
  *The dietary habits questionnaire (Kostindex) assesses dietary patterns through questions on vegetable, fruit, fish, sweets, and breakfast consumption. Scores range from 0 to 12, categorizing habits as unhealthy, moderate, or healthy to guide nutritional advice.
Change in dietary habits | At 24 months from baseline.
  To evaluate whether the intervention improves targeted lifestyle behaviors (tobacco smoking, alcohol consumption, physical activity, and dietary habits) over the 36-month period.
  Other endpoints:
  • Questionnaires Difference in the mean change in dietary habits (dietary index)* (scale 0-12).
  *The dietary habits questionnaire (Kostindex) assesses dietary patterns through questions on vegetable, fruit, fish, sweets, and breakfast consumption. Scores range from 0 to 12, categorizing habits as unhealthy, moderate, or healthy to guide nutritional advice.
Change in dietary habits | At 36 months from baseline.
  To evaluate whether the intervention improves targeted lifestyle behaviors (tobacco smoking, alcohol consumption, physical activity, and dietary habits) over the 36-month period.
  Other endpoints:
  • Questionnaires Difference in the mean change in dietary habits (dietary index)* (scale 0-12).
  *The dietary habits questionnaire (Kostindex) assesses dietary patterns through questions on vegetable, fruit, fish, sweets, and breakfast consumption. Scores range from 0 to 12, categorizing habits as unhealthy, moderate, or healthy to guide nutritional advice.
Change in physical activity | At 12 months from baseline.
  To evaluate whether the intervention improves targeted lifestyle behaviors (tobacco smoking, alcohol consumption, physical activity, and dietary habits) over the 36-month period.
  Other endpoints:
  Difference in the mean change in physical activity* (number of minutes per day).
  *The physical activity and inactivity questionnaire evaluates daily habits by measuring time spent on everyday activities, exercise, and sedentary time, including sleep.
  For physical activity:
  Higher values indicate better outcomes (more active time).
  For sedentary time:
  Higher values indicate worse outcomes (more inactive time).
Change in physical activity | At 24 months from baseline.
  To evaluate whether the intervention improves targeted lifestyle behaviors (tobacco smoking, alcohol consumption, physical activity, and dietary habits) over the 36-month period.
  Other endpoints:
  Difference in the mean change in physical activity* (number of minutes per day).
  *The physical activity and inactivity questionnaire evaluates daily habits by measuring time spent on everyday activities, exercise, and sedentary time, including sleep.
  For physical activity:
  Higher values indicate better outcomes (more active time).
  For sedentary time:
  Higher values indicate worse outcomes (more inactive time).
Change in physical activity | At 36 months from baseline.
  To evaluate whether the intervention improves targeted lifestyle behaviors (tobacco smoking, alcohol consumption, physical activity, and dietary habits) over the 36-month period.
  Other endpoints:
  Difference in the mean change in physical activity* (number of minutes per day).
  *The physical activity and inactivity questionnaire evaluates daily habits by measuring time spent on everyday activities, exercise, and sedentary time, including sleep.
  For physical activity:
  Higher values indicate better outcomes (more active time).
  For sedentary time:
  Higher values indicate worse outcomes (more inactive time).
Requirements for achieving a change in targeted lifestyle | At 12 months from baseline.
  To explore the number, type, and average time interval between intervention sessions required annually to achieve a change in the targeted lifestyle over the 36-month period.
  Other endpoint:
  • For the intervention group,
  o Effect of the number and type of lifestyle sessions with healthcare professionals on the mean change in lifestyle outcomes.
Requirements for achieving a change in targeted lifestyle | At 24 months from baseline.
  To explore the number, type, and average time interval between intervention sessions required annually to achieve a change in the targeted lifestyle over the 36-month period.
  Other endpoint:
  • For the intervention group,
  o Effect of the number and type of lifestyle sessions with healthcare professionals on the mean change in lifestyle outcomes.
Requirements for achieving a change in targeted lifestyle | At 36 months from baseline.
  To explore the number, type, and average time interval between intervention sessions required annually to achieve a change in the targeted lifestyle over the 36-month period.
  Other endpoint:
  • For the intervention group,
  o Effect of the number and type of lifestyle sessions with healthcare professionals on the mean change in lifestyle outcomes.
Effect of educational sessions | At 12 months from baseline.
  To investigate whether participation in educational sessions by participants and their relatives in the intervention group is associated with positive lifestyle changes over the 36-month period.
  Other endpoint:
  • For the intervention group,
  o Effect of participation in educational sessions (0-3 sessions) on the mean change in lifestyle outcomes.
Effect of educational sessions | At 24 months from baseline.
  To investigate whether participation in educational sessions by participants and their relatives in the intervention group is associated with positive lifestyle changes over the 36-month period.
  Other endpoint:
  • For the intervention group,
  o Effect of participation in educational sessions (0-3 sessions) on the mean change in lifestyle outcomes.
Effect of educational sessions | At 36 months from baseline.
  To investigate whether participation in educational sessions by participants and their relatives in the intervention group is associated with positive lifestyle changes over the 36-month period.
  Other endpoint:
  • For the intervention group,
  o Effect of participation in educational sessions (0-3 sessions) on the mean change in lifestyle outcomes.

CONTACTS AND LOCATIONS:
Locations (6):
- Sweden (6):
  - Psykosmottagning Centrum, Gothenburg
  - Psykosmottagning Nordost, Gothenburg
  - Psykosmottagning Öster, Gothenburg
  - Psykosmottagning Hisingen, Gothenburg
  - Psykosmottagning Väster, Gothenburg
  - Psykosmottagning Mölndal, Mölndal

IPD SHARING:
Plan to Share IPD: No
In accordance with the trial's CIP, individual participant data from this trial are not publicly available due to privacy and data protection regulations. All data are handled in compliance with the General Data Protection Regulation (EU 2016/679; GDPR) and relevant Swedish legislation, and are stored securely at Region Västra Götaland. Participants in the trial are coded with a specific record ID.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-10-21): https://cdn.clinicaltrials.gov/large-docs/01/NCT06781801/Prot_SAP_000.pdf